CLINICAL TRIAL: NCT01719224
Title: Incidence of Sleep-disordered Breathing and Upper Airway Collapsibility in Postpartum Patients and Its Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001326
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Sleep Disordered Breathing; Upper Airway Collapsibility; Upper Airway Obstruction
MeSH Terms: conditions — Sleep Apnea Syndromes; Airway Obstruction | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elevated body position (Active Comparator): We collect data about the apnea- hypopnea index, obstructive and central apneas, as well as oxygen, by comparing supine to 45 degrees elevated body position.
  Interventions: Procedure: elevated body position
- supine body position (Active Comparator): We collect data about the apnea- hypopnea index, obstructive and central apneas, as well as oxygen, by comparing supine to 45 degrees elevated body position.
  Interventions: Procedure: supine body position

INTERVENTIONS:
Procedure: elevated body position — 45 degrees elevated upper body position
  Arms: Elevated body position
Procedure: supine body position — non-elevated upper body position
  Arms: supine body position

SUMMARY:
The investigators hypothesized that sleeping in a 45 degrees elevated body position decreases the likelihood of upper airway vulnerability to collapse early after delivery. Furthermore, the investigators want to elucidate the anatomical and physiological risk factors that contribute in the upper airway obstruction in post-partum patients.

DETAILED DESCRIPTION:
After obtaining study consent, each patient underwent measurements of upper airway cross-sectional area (CSA) during daytime within 48 h after delivery. The minimum upper airway CSA was measured using acoustic pharyngometry (Eccovision Acoustic Pharyngometry; Sleep Group Solutions, Inc) in sitting, 45° elevated, and nonelevated upper body position. This method has been previously used and validated in pregnant women.

In the patients who further gave consent for the sleep study, polysomnography (PSG) was performed throughout the entire study night. Within a crossover design, patients were randomly assigned to receive first either nonelevated or 45° elevated upper body position. Position was changed after 3.5 h by a member of the team.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum mothers within 48 hours of delivery in a major academic teaching hospital.
2. Age over 18 years.
3. Admitted to the Massachusetts General Hospital OB service for the delivery.
4. Interventions will be randomly assigned to the patients enrolled in this study

Exclusion Criteria:

1. Age under 18 years.
2. History of pre-existing pulmonary and cardiac diseases, including bronchial asthma, cystic fibrosis, chronic obstructive lung disease, neck and chest tumors (thyroid, mediastinal, etc.), irradiation to the neck and/or chest, and congenital airway deformities, other critically-ill conditions.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, Ph.D, Principal Investigator — Massachusetts General Hospital Department of Anesthesia, Critical Care and Pain Medicine
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zaremba S, Mueller N, Heisig AM, Shin CH, Jung S, Leffert LR, Bateman BT, Pugsley LJ, Nagasaka Y, Duarte IM, Ecker JL, Eikermann M. Elevated upper body position improves pregnancy-related OSA without impairing sleep quality or sleep architecture early after delivery. Chest. 2015 Oct;148(4):936-944. doi: 10.1378/chest.14-2973. PMID 25905714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women during the first 48 h after delivery were included. Patients with a history of preexisting pulmonary and cardiac diseases or neck and chest tumors, as well as patients with a history of irradiation to the neck and/or chest or congenital airway deformities were not included in the study
Pre-assignment Details: 55 patients enrolled in the study and all of them successfully completed acoustic pharyngometry during wakefulness. 36 of 55 participants were randomized to receive one of the two sleeping positions first. Of those not randomized, 19 declined to participate in the overnight PSG recording.
Groups:
- Experimental: Elevated Position, Then Non-Elevated Position: In the beginning of the study night, participants were placed in a sleeping position at 45 degrees upper body elevation. After 3.5h, a study member changed the patients bed to a non-elevated position. We collected data about the apnea- hypopnea index, obstructive and central apneas, as well as oxygen during the study night.
- Experimental: Non-Elevated Position, Then Elevated Position: In the beginning of the study night, participants were placed in a non-elevated sleeping position. After 3.5h, a study member changed the patients bed to a 45 degrees upper body position. We collected data about the apnea- hypopnea index, obstructive and central apneas, as well as oxygen during the study night.
Period: Intervention 1: Sleeping Position 1
Arm/Group | Experimental: Elevated Position, Then Non-Elevated Position | Experimental: Non-Elevated Position, Then Elevated Position
Started | 18 | 18
Completed | 14 | 16
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Intervention 2: Position Change(At 3.5h)
Arm/Group | Experimental: Elevated Position, Then Non-Elevated Position | Experimental: Non-Elevated Position, Then Elevated Position
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 55 patients enrolled in the study and all of them successfully completed acoustic pharyngometry during wakefulness. 36 of 55 participants were randomized to receive one of the two sleeping positions first. Of those not randomized, 19 declined to participate in the overnight PSG recording.
Groups:
- Total Study Population (N=55): Fifty-five patients were enrolled within 48 hours after delivery from two newborn family units at MGH hospital.
Arm/Group | Total Study Population (N=55)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.13 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
BMI prior to pregnancy [Mean (Standard Deviation); unit: kg/m^2] | 25.82 (6.8)
BMI end of pregnancy [Mean (Standard Deviation); unit: kg/m²] | 30.84 (7)
Delivery method: C-Section [Number; unit: participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI), Defined as the Number of Apneas and Hypopneas Per Hour of Sleep
Description: We conduct polysomnography in non-elevated and 45 degrees elevated body position, to show the effect of body position in context of sleep disordered breathing.We collect data of the apnea-hypopnea-index, central apneas, obstructive apneas and oxygen.
Time Frame: 48 hours after delivery
Population: 55 women (older than 18 years) were recruited within 48 h after delivery. Polysomnography (PSG) was performed throughout the entire study night. Within a crossover design, patients were randomly assigned to receive first either nonelevated or 45° elevated upper body position. Position was changed after 3.5 h by a member of the team.
Measure: Mean (Standard Error); unit: Apneas and hypopneas per hour of sleep
Groups:
- Elevated Upper Body Position: We collect data about the apnea- hypopnea index, obstructive and central apneas, as well as oxygen, by comparing supine to 45 degrees elevated body position.
  elevated body position: 45 degrees elevated upper body position
- Non-elevated Upper Body Position: We collected data about the apnea- hypopnea index, obstructive and central apneas, as well as oxygen, by comparing supine to 45 degrees elevated body position.
  Supine body position: non-elevated upper body position
Arm/Group | Elevated Upper Body Position | Non-elevated Upper Body Position
Number analyzed (Participants) | 34 | 32
Apneas and hypopneas per hour of sleep | 4.5 (1.4) | 7.7 (2.2)

2. Secondary Outcome: Minimum Upper Airway Cross-sectional Area: to Elucidate the Anatomical and Physiological Risk Factors That Contribute to the Upper Airway Obstruction in Post-partum Patients
Description: Each patient underwent measurements of upper airway CSA during daytime within 48 h after delivery. The minimum upper airway CSA was measured using acoustic pharyngometry (Eccovision Acoustic Pharyngometry; Sleep Group Solutions, Inc) in sitting, 45° elevated, and nonelevated upper body position.
Time Frame: 48 hours after delivery
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- Sitting Position: Fifty-five patients were enrolled within 48 hours after delivery, and all of them successfully completed acoustic pharyngometry during wakefulness. Each patient had the pharyngemtry measurements in a sitting position
- Non-elevated Position; 45 Degree Elevation: Fifty-five patients were enrolled within 48 hours after delivery, and all of them successfully completed acoustic pharyngometry during wakefulness. Each patient had the pharyngemtry measurements in a non-elevated (supine) position.
Arm/Group | Sitting Position | Non-elevated Position | 45 Degree Elevation
Number analyzed (Participants) | 55 | 55 | 55
cm^2 | 1.54 (0.1) | 1.35 (0.1) | 1.46 (0.1)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Elevated Body Position | Supine Body Position
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations include the fact that we report single-center-data and the inability draw conclusions on long-term outcome due to cross-over study-design.

No direct implications on sleep-apnea during pregnancy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No